CLINICAL TRIAL: NCT05913115
Title: A Phase 1 Open-Label, Dose-Finding Study Evaluating Safety and Pharmacokinetics of FPA144 in Japanese Patients With Advanced Gastric or Gastroesophageal Cancer
Brief Title: A Study Evaluating Safety and Pharmacokinetics of FPA144 in Japanese Patients With Advanced Gastric or Gastroesophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FPA144-002
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Gastric or Gastroesophageal Cancer
Keywords: FPA144
MeSH Terms: interventions — bemarituzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FPA144 (Experimental): Participants will receive escalating doses of FPA144. On completion of Cycle 1 (Cycles = 28 days in length) participants may participate in an optional Extended Treatment Period based on the Investigator's discretion, which begins on Day 1 of Cycle 2. FPA144 will be administered once every 2 weeks (Q2W) in 4-week cycles until disease progression, or until the patient meets any of the other withdrawal criteria.
  Interventions: Drug: FPA144

INTERVENTIONS:
Drug: FPA144 — FPA144 will be administered intravenously Q2W.
  Other Names: Bemarituzumab

SUMMARY:
The main objectives of this study are:

* To determine the recommended dose (RD) of FPA144 in participants with gastric or gastroesophageal cancer (hereafter referred to as gastric cancer)
* To evaluate the safety of escalating doses of FPA144 in participants with gastric cancer
* To characterize the pharmacokinetic (PK) profile of single and multiple doses of intravenously administered FPA144 in participants with gastric cancer

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma that is locally recurrent or metastatic and has progressed following standard treatment or is not appropriate for standard treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate hematological, liver and kidney function. Measurable or non-measurable disease
* Archival tumor tissue for determination of FGFR2 status

Key Exclusion Criteria:

* Untreated or symptomatic central nervous system (CNS) metastases
* Clinically significant cardiac disease
* Peripheral sensory neuropathy >/= Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Active infection requiring systemic treatment
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known active or chronic hepatitis B or C infection
* Prior treatment with any selective inhibitor of the fibroblast growth factor (FGF)-FGFR pathway
* Known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
* Known positivity for human epidermal growth factor receptor 2 (HER2)
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience Grade 3 or Grade 4 Dose-limiting Toxicities (DLTs) | Day 1 to Day 28 of Cycle 1
  DLTs are defined as specific adverse events (AEs) or clinically laboratory abnormalities that occur during the DLT observation period (Day 1 to Day 28 of Cycle 1; cycle = 28 days), that the Cohort Review Committee (CRC) assess as related to FPA144. Events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03:
  * Grade 3: Severe or medically significant but non-immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; severe AE
  * Grade 4: Life-threatening consequences; urgent intervention indicated
Area Under Serum Concentration-time Curve (AUC) of FPA144 | Cycle 1: Pre-dose (within 4 hours prior to infusion on Day 1) and 0.5, 3, 6, 24, 72, and 168 hours after end of infusion; Subsequent cycles: Pre-dose (within 4 hours prior to infusion) and 0.5 hours after end of infusion on Day 1 and Day 15
Maximum Serum Concentration (Cmax) of FPA144 | Cycle 1: Pre-dose (within 4 hours prior to infusion on Day 1) and 0.5, 3, 6, 24, 72, and 168 hours after end of infusion; Subsequent cycles: Pre-dose (within 4 hours prior to infusion) and 0.5 hours after end of infusion on Day 1 and Day 15
Trough Serum Concentration (Ctrough) of FPA144 | Cycle 1: Pre-dose (within 4 hours prior to infusion on Day 1) and 0.5, 3, 6, 24, 72, and 168 hours after end of infusion; Subsequent cycles: Pre-dose (within 4 hours prior to infusion) and 0.5 hours after end of infusion on Day 1 and Day 15
Clearance (CL) of FPA144 | Cycle 1: Pre-dose (within 4 hours prior to infusion on Day 1) and 0.5, 3, 6, 24, 72, and 168 hours after end of infusion; Subsequent cycles: Pre-dose (within 4 hours prior to infusion) and 0.5 hours after end of infusion on Day 1 and Day 15
Terminal Half-life (t1/2) of FPA144 | Cycle 1: Pre-dose (within 4 hours prior to infusion on Day 1) and 0.5, 3, 6, 24, 72, and 168 hours after end of infusion; Subsequent cycles: Pre-dose (within 4 hours prior to infusion) and 0.5 hours after end of infusion on Day 1 and Day 15
Volume of Distribution of FPA144 | Cycle 1: Pre-dose (within 4 hours prior to infusion on Day 1) and 0.5, 3, 6, 24, 72, and 168 hours after end of infusion; Subsequent cycles: Pre-dose (within 4 hours prior to infusion) and 0.5 hours after end of infusion on Day 1 and Day 15

SECONDARY OUTCOMES:
Number of Participants who Experience Treatment-emergent AEs (TEAEs) | Approximately 1 year
  TEAEs will be graded using the NCI CTCAE version 4.03. Any clinically significant laboratory abnormalities will also be reported as TEAEs.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- Japan (2):
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com